CLINICAL TRIAL: NCT05519709
Title: Investigation of Scapular Dyskinesia, Shoulder Mobilization and Serve Speed Variables in Asymptomatic Adolescent Tennis Players
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Irem Kurt, Physiotherapist, Lecturer, Istanbul University - Cerrahpasa
Other Study IDs: IUC-IGU
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Tennis; Adolescent; Scapular Dyskinesia; Shoulder Mobilization; Serve Speed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asymptomatic Adolescent Tennis Players: Adolescent tennis players aged 7-17 years who have been actively attending tennis club for at least 1 year will be form adolescent tennis players groups. The age, body weight (kg) and height (centimeter) of each individual included in the study will record. The assessment form, which includes demographic data such as, training duration(min/day), frequency (times/week) and sport age will record by asking the parents. All measurements will be take before lesson and without warm-up. All measurements will be evaluate by an experienced physiotherapist.

SUMMARY:
Tennis is a sport where high performance, strokes and wide ranges of motion around the court must be created and high-strength movements are repeated repeatedly. Speed and control are important in terms of sportive performance during the serve throw in tennis. While these actions are taking place, a dynamic load that exceeds the physiological limits of the joint is placed on the shoulder. Disruption in the kinetic chain can cause injury to the shoulder. In this regard, the incidence of tennis injuries is approximately 21.5 injuries per 1000 training hours. The glenohumeral joint creates a wide range of motion for the shoulder and is also biomechanically related to the scapula. Scapular dyskinesia, the pathological position of the scapula, has been associated with common pathologies such as rotator cuff tears, labral tears, and shoulder impingement. Although there are studies with different opinions about the causality of scapular dyskinesia, the current literature has reported that scapular dyskinesia is indirectly associated with shoulder pain in overhead athletes. Achieving maximum shoulder performance in sports that require overhead activities such as tennis largely depends on the delicate balance between the scapula and the clavicle, humerus and rib cage joints. Tennis, which is an increasingly widespread sport in our country, exposes the shoulder joints to high stresses. If changes are not detected and necessary precautions are not taken, the shoulder structure may be at risk of injury. In the current literature review, no study was found that evaluated the relationship between scapular dyskinesia, shoulder mobility and serving speed in tennis players. The aim of our study is to evaluate the effects of scapular dyskinesia, glenohumeral joint mobility and posterior capsule tension on serving speed in tennis players. It is thought that the results to be obtained from our study will guide the creation of appropriate exercise programs in athlete training by determining the effects on sportive performance by determining the changes seen or to be seen in the shoulder complexes of tennis athletes.

ELIGIBILITY:
Inclusion Criteria:

* 12-20 ages
* Volunteer
* Does not have any cognitive, mental and psychological problems,
* Does not have any systemic diseases such as rheumatoid arthritis,
* Does not have any neurological problems,
* Additionally, the criteria for the tennis players included more than 1 years of tennis experience.

Exclusion Criteria:

* Having severe neurological, visual and auditory problems that may prevent the application of assessment parameters
* Children and their families who cannot obtain written consent from their families.
* Having communication problems

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Asymtomatic dolescent tennis players aged 7-17 years who have been actively attending a tennis club for at least 1 year will be form tennis players group.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Shoulder Protraction | Baseline
  Shoulders in protraction; It will be determined by the distance of the posterior corner of the lateral acromion process from the bed to 2.5 cm or more. In order to prevent measurement changes due to humeral rotation, the person will be positioned on the abdomen with the elbow flexed, with the shoulder in a neutral position. The measurement with the caliper will be recorded in cm. The inter-rater reliability of the test was good and the intra-class correlation coefficient was found to be ICC> 0.90.
Pectoralis Minor Length Measurement | Baseline
  The subject standing upright, with the arm to be tested relaxed, the distance between the origin and insertion of the muscle will be measured in cm with a caliper as linear length. The origin of the muscle is defined as the inferior part of the 4th rib, one finger lateral to the sternocostal junction, and the insertion site is the medio-inferior part of the coracoid process. Multiplying the longitudinal part of the individual by 100 of the distance between the origin and insertion gives the pectoralis minor index (PMI). The PMI allows each measurement to be normalized to the subject's height so that the individual's relative pectoralis minor length at rest is obtained. It was determined that the pectoralis minor length measurement had good inter-rater reliability (ICC: 0.85) and showed good validity (ICC = 0.96) when compared with the 3D electromagnetic system. Its reliability among evaluators varies between 0.53-0.56.
Passive Shoulder Internal Rotation (IR) and External Rotation (ER) Mobility Flexibility Measurement | Baseline
  Passive IR and ER joint range of motion measurements of the individual will be made with a goniometer. While the individual is lying in the supine position, the measurement will be performed in degrees (°) by taking the shoulder joint to 90° abduction, the elbow joint to 90° flexion and the forearm to neutral. During passive IR assessment, measurement will be stopped when the postero-lateral of the acromion is lifted off the ground to prevent scapular movements with visual control. The intra-rater reliability (ICC) for IR ranged from 0.38 to 0.60 and for ER to range from 0.78 to 0.88.
Active Shoulder IR and ER Mobility Flexibility Measurement | Baseline
  For active IR and ER mobility (flexibility) measurement, cervical vertebral spinous process (C7) and 5th thoracic vertebra spinous process (T5) will be determined as reference points. The distance between the thumb and C7 will be measured in cm with a tape measure, by asking the individual to make maximum external rotation by bringing the arm behind the neck with the thumb pointing down. Then, the individual will be asked to bring the arm behind the waist to maximum internal rotation with the thumb pointing up, and the distance between the tip of the thumb and the T5 will be measured in cm with a tape measure. It was stated that the reliability of the IR flexibility measurement was 0.44, the reliability of the ER flexibility measurement was 0.39, and both measurements were reliable.
Shoulder Posterior Tension Test | Baseline
  It will be done while the person is in the side-lying position. With the subject's humerus in a neutral position, the arm will be abducted 90° and the elbow flexed to 90°, while the evaluator will stabilize the scapula in a fully retracted position while the arm will be passively pulled down into horizontal adduction. At the final destination, the distance between the bed and the medial epicondyle will be measured in cm and recorded. The same measurement will be repeated for the other shoulder and recorded.
Scapular Dyskinesia- Lateral Scapular Slide Test | Baseline
  The Lateral Scapular Slide Test (LSST), designed by KIBLER in 1991, was used to evaluate scapular dyskinesia. The test includes three positions with the arms at the sides in a neutral position, the hands at the waist, the thumbs pointing back, and the shoulders at 90° abduction and the arms in maximum internal rotation. In all 3 positions, the distance between the lower angle of the scapula and the spinous process of the nearest thoracic vertebra will be measured bilaterally with a caliper and recorded in cm. A bilateral scapular distance greater than 1.5 cm will be recorded as the presence of scapular dyskinesia. The LSST is a test that can be used clinically, and its test-retest reliability can vary between 0.43 and 0.88, and its inter-rater reliability can vary between 0.75 and 0.85.
Scapular Retraction Test | Baseline
  For the Scapular Retraction Test (SRT), the participant will be positioned with their back to the researcher. The investigator will stand next to the participant, stabilizing the scapula in retraction. The test will be considered positive if pain occurs when the scapula is stabilized in retraction.
Scapular Support Test | Baseline
  While the participant is doing active shoulder flexion, an upward rotation movement will be applied to the researcher participant's scapula. The test will be considered positive if the shoulder arc of motion increases or the pain in the painful arch decreases/passes when the investigator rotates the scapula upwards.
Measuring Service Speed | Baseline
  Radar gun will be used while measuring service speed. Athletes will perform upper extremity mobility and warm-up for 5 minutes in order to reach the maximum level of service speed, and then serve 2 sets of 8 reps. Athletes will throw tennis balls 1 m away from the center service line, using their own rackets and in accordance with the standards of the International Tennis Federation 6-7. cm in diameter, weighing 58.4 g) will serve. The radar gun will be located 4 m behind the center of the baseline at an altitude of approximately 2.2 m. The gun velocity will be evaluated in kilometers per hour with a calibrated radar gun (Bushnell 1101911 Velocity Speed Gun). Athletes will be asked to serve with 8 maximal repetitions. The average of the services with the maximum speed will be used. There is a 30 s rest period between service shots. Its reliability has been proven with ICC values ranging from 0.91-0.94.

SECONDARY OUTCOMES:
Upper Extremity Physical Function Measurement | Baseline
  Quick-Disabilities of the Arm, Shoulder and Hand (Q-DASH) will be used to measure upper extremity physical function. The questionnaire includes 11 titles extracted from the long version and each question consists of a 5-point scale. Total score is calculated with the formula [(sum of n answers) /n-1] ×25, n= indicates the total number of questions answered. The total score ranges from 0 (no disability) to 100 (severe disability). 0- 15: 'no problem', 16-40: 'there is a problem but can work', 40 and above: 'not able to work'.

CONTACTS AND LOCATIONS:
Locations (1):
- İrem Kurt, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided